CLINICAL TRIAL: NCT00315952
Title: Open-Label Randomized Two-Way Crossover Pilot Study to Estimate the Effects of Inhaled vs. IV Infusion of Human Insulin With Regards to Glucose Disposal in Subjects With Type 1 Diabetes Mellitus
Brief Title: Study to Estimate the Effects of Inhaled Versus Intravenous (IV) Infusion of Human Insulin in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 06020777
Record Dates: First submitted 2006-04-17; First posted 2006-04-19 (Estimated); Last update posted 2008-02-18 (Estimated); Status verified 2008-02

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: type 1 diabetes mellitus; inhaled insulin; Positron Emission Tomography
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Exubera

INTERVENTIONS:
Drug: Exubera

SUMMARY:
University of Pittsburgh Medical Center (UPMC) diabetes research physicians are studying the action in muscle tissue of "inhaled" insulin (Exubera®) and "infused" (intravenous or IV) insulin on blood sugar control in people with type 1 diabetes. Type 1 diabetics often take 2-4 shots of insulin every day. Exubera may offer an alternative to these insulin injections.

DETAILED DESCRIPTION:
A dry powder insulin formulation delivered by an aerosol inhaler has been in clinical development for use in types 1 and 2 diabetes mellitus (DM) and just recently (1-27-06) received approval from the U.S. Food and Drug Administration (FDA) for the clinical treatment of diabetes. Administration of insulin without the need for subcutaneous (SC) injection is an attractive alternative for patients with diabetes. There are preclinical and clinical data that indicate inhalation of insulin results in a more potent effect on glucose disposal and a lower fasting glucose than is attained with equivalent dosing of SC or intravenous (IV) insulin. The physiological mechanism(s) are unclear, but occur even when matched for pharmacokinetics.

The current proposal seeks primarily to more fully delineate whether there are physiological differences in the metabolic effects of inhaled compared to IV infused insulin, giving IV insulin to match the pharmacokinetics (PK) achieved with inhaled insulin.

There are 3 specific aims:

1. The first aim is to establish a protocol for matching the PK of inhaled insulin with the PK of intravenously infused insulin. An infusion algorithm has been developed and will be tested and refined in healthy volunteers (n = 3-5), and will be used for the physiological studies (aims) outlined below.
2. The second aim is to perform Positron Emission Tomography (PET) imaging of [18F]-FDG uptake by muscle, following administration of a single dose of inhaled compared to infused insulin. Volunteers with type 1 DM (n =12) will be studied, serving as his/her within-subject control, under each condition of insulin administration.

   In these type 1 diabetes mellitus (type 1 DM) volunteers, we will test the hypothesis that a single dose of inhaled versus infused insulin, matched for arterial concentrations, causes greater stimulation of muscle glucose uptake.
3. The third aim is to determine overnight rates of glucose production and plasma glucose after a single pre-dinner dose of inhaled compared to IV infused insulin. The same 12 volunteers studied for Aim 2 will be studied the evening preceding the PET imaging studies and will serve as his/her within-subject control, under each condition of insulin administration.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 50 years old
* Body mass index (BMI) 20 to 27 kg/m2 and a total body weight > 50 kg (110 lbs)
* Blood pressure: systolic < 150; diastolic < 95.
* Type 1 DM
* Have diagnosed diabetes type 1 for a minimum of 12 months prior to study entry
* In good general health with no evidence or history of clinically significant hematological, renal, endocrine (other than diabetes), pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing)
* Hematocrit (Hct) > 34%
* ALT < 60; AST < 60
* Alkaline phosphatase (Alk Phos) < 150
* Sensitive thyroid-stimulating hormone (sTSH) < 6
* Fasting (morning) glucose 100-160 mg/dl
* Documented hemoglobin A1c (HbA1c) < 7.5% at time of entry
* Triglycerides < 175
* Cholesterol < 275

Exclusion Criteria:

* Exclude if unable to master use of the inhalation device after 3 attempts
* Exclude if positive urine drug screen
* Exclude if any episodes of severe hypoglycemia in the past 3 months
* Exclude if pregnant or breastfeeding or unwilling to use an acceptable method of non-hormonal contraception from at least 14 days prior to the first dose of Exubera® until study is completed.
* Exclude if any history of (h/o) asthma or chronic obstructive pulmonary disease (COPD)
* Exclude if forced expiratory volume in one second (FEV1) or forced vital capacity (FVC) < 70% predicted
* Exclude if treatment with an investigational drug within 30 days preceding the first dose of trial medication.
* Exclude if blood donation of approximately 1 pint (500 mL) within 56 days prior to dosing
* Exclude if unable or unwilling to comply with the protocol as written
* Exclude if any use of tobacco or nicotine containing products within the past 6 months
* Exclude if history of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for men (1 drink = 5 ounces of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months of screening
* Exclude if claustrophobic, any surgical or vascular implants or pacemakers, or any metal in the body

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2006-04; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To perform positron emission tomography (PET) imaging of [18F]-fluoro-deoxy-glucose (FDG) uptake by muscle, following administration of a single dose of inhaled compared to infused insulin in volunteers with type 1 diabetes

SECONDARY OUTCOMES:
To determine overnight rates of glucose production and plasma glucose after a single pre-dinner dose of inhaled compared to IV infused insulin in volunteers with type 1 diabetes

CONTACTS AND LOCATIONS:
Overall Officials: David E. Kelley, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States